CLINICAL TRIAL: NCT00412295
Title: Evaluation of Alcon Ladarvision Wavefront-Guided PRK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources and not because of any concern with the safety or effectiveness of the procedures studied.
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Samantha B. Rodgers, MD, PRS Account holder, Walter Reed Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU#04-23006
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2014-12

CONDITIONS: Myopia
Keywords: Naturally occuring myopia with or without astigmatism.; Wavefront errors
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Wavefront-guided PRK
  Interventions: Device: Alcon Ladarvision (Wavefront-guided PRK)

INTERVENTIONS:
Device: Alcon Ladarvision (Wavefront-guided PRK) — Wavefront-guided PRK using Alcon Ladarvision

SUMMARY:
The purpose of this study is to:

1. determine the safety of wavefront guided PRK
2. evaluate the efficacy of wavefront guided PRK
3. evaluate the differences in visual quality after treatment of wavefront guided PRK

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from those active duty soldiers that have requested refractive surgery. Subjects must be eligible for medical care at WRAMC.
* Male or female, of any race, and at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
* Manifest refractive spherical equivalent (MSE) of up to -6 diopters (D) at the spectacle plane with refractive cylinder up to 3.00D.
* At least five images must be capturesd in both eyes (dilated) with a pupil size of at least 7mm.
* Manifest refraction and LADARWave™ refractions must be within 1.00 D and the CustomCornea® software must allow for treatment with a 6.5mm minor axis and 9mm ablation zone.
* Best spectacle corrected visual acuity of 20/20 or better in both eyes.
* Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12-month period immediately preceding the baseline examination, sa confirmed by clinical records.
* Soft contact lens users must have removed their lenses at least 2 weeks before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least 4 weeks prior to baseline measurements adn have 2 central Keratometry readings and 2 manifest refractions taken at least 1 week apart that do not differ by more than 0.50D in either meridian; mires should be regular.
* Located it the greater Washington DC Area for a 12-month period.
* Exhibits strong motivation for attending the follow-up visits.
* Consent of the subject's command (active duty) to participate in the study.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Female subjects who are pregnant, breast feeding or intend to become pregnant during the study.
* Concurrent topical or systemic medications that may impair healing, including corticosteriods, antimetabolites, isotretinoin, amiodarone hydrochloride and/ or sumatripin.
* Medical condition(s), which, in the judgement of the investigator, may impair healing, including but not limited to: collagen vascular diseases and ocular herpes zoster or simplex.
* Active ophthalmic disease, neovascularization of the cornea within 1mm of the intended ablation zone, or clinically significant lens opacity.
* Evidence of glaucoma or an intraocular pressure greater than 22mm Hg at baseline.
* Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
* History of recurrent erosions or epithelial baewsment dystrophy.
* Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
* Any physical or mental impairment that would preclude participation in any of the examinations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity (CDVA) | 12 months
  CDVA (logMAR unit and/or snellen equivalent) will be measured to determine safety of wavefront guided PRK.
Uncorrected distance visual acuity (UDVA) | 12 months
  UDVA (logMAR unit and/or snellen equivalent) will be measured to determine effectiveness of wavefront guided PRK.

CONTACTS AND LOCATIONS:
Overall Officials: STEVEN SCHALLHORN, MD, Principal Investigator — United States Naval Medical Center, San Diego; KRAIG S BOWER, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - Naval Medical Center, San Diego, California
  - Walter Reed Army Medical Center, Center For Refractive Surgery, Washington D.C., District of Columbia